CLINICAL TRIAL: NCT06488768
Title: Duration of Peripheral Nerve Blocks in Opioid Tolerant Individuals - A Volunteer Blinded Matched Case-control Study
Acronym: OPITOBLOK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charlotte Runge (Other)
Responsible Party: Sponsor-Investigator, Charlotte Runge, Senior Consultant, Regionshospitalet Silkeborg
Organization: Regionshospitalet Silkeborg (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-509351-13-00
Record Dates: First submitted 2024-06-17; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Nerve Block; Opioid Tolerance
Keywords: Nerve Block; Opioid tolerance; Radialis Nerve block

STUDY DESIGN:
Intervention Model Description: A volunteer blinded matched case-control study.
Who Masked: Investigator
Masking Description: An investigator blinded to the volunteer's opioid status will perform all the sensory and motor tests after thorough instruction in this procedure. Only the primary investigator will have the knowledge of opioid status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid tolerant (Experimental): Daily use of opioid of 60 mg or more
  Interventions: Other: Radial nerve block
- Opioid naive (Experimental): No use of opioids within the last 30 days
  Interventions: Other: Radial nerve block

INTERVENTIONS:
Other: Radial nerve block — Ultrasound-guided Radial nerve block. Conducted with 10 mL of Lidocaine 2%. Ultrasound image are stored for documentation.

SUMMARY:
Do peripheral nerve blocks work shorter if you are on opioids?

Background:

Peripheral nerve blocks effectively alleviate postoperative pain. Animal studies and human research indicate that opioid tolerance results in reduced effectiveness of local analgesics. This applies to both central nerve blockade and infiltration anaesthesia. The impact on peripheral nerve block in humans has not been evaluated. The aim of the study is to assess the onset time and duration of a radial nerve block in opioid tolerant individuals compared to opioid naive individuals. We hypothesise that peripheral nerve blocks cause shorter sensory and motor block in opioid-tolerant compared to opioid-naive counterparts.

Methods:

Twenty opioid-tolerant individuals will be matched by sex and age with opioid-naïve counterparts. Participants will undergo an ultrasound-guided radial nerve block. The onset time and duration of motor and sensory blockade will be tested and measured. The primary outcome is difference in duration of sensory nerve blockade between the two groups. The secondary outcomes include the onset time of sensory blockade, onset time of motor blockade, and difference in duration of motor nerve blockade.

Perspectives:

The data from this study will provide evidence for the duration of peripheral nerve block in opioid tolerant individuals and support if a specific postoperative protocol for opioid tolerant individuals is needed or it should be of special attention.

ELIGIBILITY:
Inclusion criteria for opioid group

* Age > 18 years old
* ASA 1-3
* Chronic pain, defined as persisting pain for more than three months
* Daily use of more than 60 mg of morphine equivalent in more than 7 days
* Legally competent and able to give informed consent

Inclusion criteria for the opioid naive control group

* Age > 18 years old
* ASA 1-3
* No use of opioids within 30 days prior to participation
* Legally competent and able to give informed consent

Exclusion Criteria:

* Age > 84 years old
* Volunteers who cannot cooperate with the study
* Volunteers who cannot understand or speak Danish
* Allergy to the lidocaine or the preservatives used in the study
* Alcohol or drug abuse other than opioids
* Peripheral neuropathy at the upper limb non-dominant arm
* Pathology or previous major surgery to the upper limb
* Active signs of infection in the cutaneous area of injection
* Pregnancy at the time of the trial
* Partial or complete 2nd or 3rd degree atrioventricular heart block without a pacemaker
* Severe liver disease
* Severe kidney disease and reduced kidney function (eGFR below 30 mL/min)
* Daily treatment with drugs that are structurally related to local analgesics or class IB antiarrhythmics, as the toxic effects are additive
* Daily treatment with class III antiarrhythmics e.g., amiodarone.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the duration of sensory block for a radial nerve block between opioid-tolerant and opioid-naive individuals. | Up to one hour after nerve block placement.
  Following the injection of local anaesthetic, motor and sensory assessments will be conducted at 30-second intervals until complete sensory and motor blockade, respectively. These assessments will involve comparisons with the contralateral side.
  Sensory testing will be performed on the dorsal side of the 1. intermetacarpal area (the space between the thumb and the index finger) and the proximal dorsolateral area of the antebrachium. In both areas seeking to explore the boundaries of the innervation area.
  Dual testing is performed to accommodate interindividual variabilities in dermatomes. Sensation will be evaluated with a monofilament (Touch Test, 60 g; Stoelting, Co, Wood Dale, IL) using a 11-point sensory scale:
  5 = extremely intense sensation 0 = normal sensation.
  -5 = no sensation.

SECONDARY OUTCOMES:
The difference in the onset time of sensory block from a radial nerve block between opioid-tolerant and opioid-naive individuals. | Up to one hour after nerve block placement.
  Following the injection of local anaesthetic, motor and sensory assessments will be conducted at 30-second intervals until complete sensory and motor blockade, respectively. These assessments will involve comparisons with the contralateral side.
  Sensory testing will be performed on the dorsal side of the 1. intermetacarpal area (the space between the thumb and the index finger) and the proximal dorsolateral area of the antebrachium. In both areas seeking to explore the boundaries of the innervation area.
  Dual testing is performed to accommodate interindividual variabilities in dermatomes. Sensation will be evaluated with a monofilament (Touch Test, 60 g; Stoelting, Co, Wood Dale, IL) using a 11-point sensory scale:
  5 = extremely intense sensation 0 = normal sensation.
  -5 = no sensation.
The difference in the onset time of motor block from a radial nerve block between opioid-tolerant and opioid-naive individuals. | Up to one hour after nerve block placement.
  Following the injection of local anaesthetic, motor and sensory assessments will be conducted at 30-second intervals until complete sensory and motor blockade, respectively. These assessments will involve comparisons with the contralateral side.
  With the arm placed in pronated position on a flat and solid surface the ability to dorsally flex the wrist is used to evaluate motor block on a Modified Bromage three-point scale: 0 = normal contraction.
  * 1 = reduced contraction.
  * 2 = no contraction.
The difference in the duration of motor block for a radial nerve block between opioid-tolerant and opioid-naive individuals. | Up to one hour after nerve block placement.
  Following the injection of local anaesthetic, motor and sensory assessments will be conducted at 30-second intervals until complete sensory and motor blockade, respectively. These assessments will involve comparisons with the contralateral side.
  With the arm placed in pronated position on a flat and solid surface the ability to dorsally flex the wrist is used to evaluate motor block on a Modified Bromage three-point scale: 0 = normal contraction.
  * 1 = reduced contraction.
  * 2 = no contraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: Within one year of the end of the trial.